CLINICAL TRIAL: NCT05082896
Title: Multicentre ObseRvational Study in Posterior mecHanical thrombEctomy: conscioUs Sedation vs General aneSthesia: MORPHEUS STROKE REGISTRY
Brief Title: Multicentre ObseRvational Study in Posterior mecHanical thrombEctomy: conscioUs Sedation vs General aneSthesia
Status: Completed | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor
Other Study IDs: MORPHEUS STROKE REGISTRY
Record Dates: First submitted 2021-09-13; First posted 2021-10-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Thrombectomy; General Anesthesia; Conscious Sedation; Posterior Circulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conscious Sedation
  Interventions: Procedure: Type of anesthesia choice
- General Anesthesia
  Interventions: Procedure: Type of anesthesia choice

INTERVENTIONS:
Procedure: Type of anesthesia choice — Use of conscious sedation vs. general anesthesia

SUMMARY:
The association of conscious sedation vs. general anesthesia in ischemic stroke with posterior circulation occlusions undergoing endovascular therapy, is istill unknown.

No prospective or clinical trials have studied this effect on posterior circulation strokes.

The choice of anesthetic regimen is ussually depending on local stroke-team protocols or neurointerventional preference.

MORPHEUS Stroke Registry is a prospective multicentre observational study that investigates the association between anestheisa and functional outcome in patients with posterior circulation large vessel occlusion treated endovascularly.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years
* Evidence of posterior arterial occlussion (basilar artery, intracranial vertebral artery and posterior cerebral artery)
* Patients eligible for mechanical thrombectomy

Exclusion Criteria:

* Patient's refusal to participate
* Arterial recanalization prior to endovascular thrombectomy attempt
* Patient unable to present or be available for follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients eligible for mechanical thrombectomy due to ischemic stroke and presence of arterial occlusion in intracranial posterior circulation
Sampling Method: Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Functional independence at 3 months | 3 months
  Rate of functional independence (modified Rankin Scale 0-2) at 3 months

SECONDARY OUTCOMES:
First Pass Effect | 1 day
  Rate of complete successful recanalization (mTICI 2c-3) with one single pass of device
Mortality | 3 months
  Rate of mortality at 3 months
Successfull recanalization and complete recanalization according to endovascular technique | 1 day, revascularization grade will be assessed
  Rate of mTICI 3 and mTICI 2b-3 according to endovascular technique (contact aspiration, stentriever or combined)
Number of passes | 1 day, number of device passes will be assessed
  Number of intracranial thrombectomy passes to achieve final reperfusion
NIHSS at 24 hours | 24 hours
  Rate of neurological status at 24 hours, dramatical neurological improvement after mechanical thrombectomy
Type of anesthesic and outcome | 3 months
  Study of the type of anesthesic choice and complications, time of intubation and
Length of stentretriever and recanalization | 1 day, stentretriever type will be assessed
  Rates of FPE and succesful recanalization according to the length of stentretriever used
Arterial hypotension during anesthesic induction and outcome | 3 months
  Study of arterial hypotension during anesthesic induction and outcome
Bridging therapy and neurologial/functional outcomes | 1 day, type of previous fibrinolytic use will be assessed
  To study the association between bridging therapy and reperfussion rates, neurological status and funtional independence at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Doctor Josep Trueta de Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Hu G, Shi Z, Li B, Shao W, Xu B. General anesthesia versus monitored anesthesia care during endovascular therapy for vertebrobasilar stroke. Am J Transl Res. 2021 Mar 15;13(3):1558-1567. eCollection 2021. PMID 33841679
- [Result] Wu L, Jadhav AP, Chen J, Sun C, Ji K, Li W, Zhao W, Li C, Wu C, Wu D, Ji X. Local anesthesia vs general anesthesia during endovascular therapy for acute posterior circulation stroke. J Neurol Sci. 2020 Sep 15;416:117045. doi: 10.1016/j.jns.2020.117045. Epub 2020 Jul 16. PMID 32717535
- [Result] Jadhav AP, Bouslama M, Aghaebrahim A, Rebello LC, Starr MT, Haussen DC, Ranginani M, Whalin MK, Jovin TG, Nogueira RG. Monitored Anesthesia Care vs Intubation for Vertebrobasilar Stroke Endovascular Therapy. JAMA Neurol. 2017 Jun 1;74(6):704-709. doi: 10.1001/jamaneurol.2017.0192. PMID 28395002
- [Result] Campbell BCV, van Zwam WH, Goyal M, Menon BK, Dippel DWJ, Demchuk AM, Bracard S, White P, Davalos A, Majoie CBLM, van der Lugt A, Ford GA, de la Ossa NP, Kelly M, Bourcier R, Donnan GA, Roos YBWEM, Bang OY, Nogueira RG, Devlin TG, van den Berg LA, Clarencon F, Burns P, Carpenter J, Berkhemer OA, Yavagal DR, Pereira VM, Ducrocq X, Dixit A, Quesada H, Epstein J, Davis SM, Jansen O, Rubiera M, Urra X, Micard E, Lingsma HF, Naggara O, Brown S, Guillemin F, Muir KW, van Oostenbrugge RJ, Saver JL, Jovin TG, Hill MD, Mitchell PJ; HERMES collaborators. Effect of general anaesthesia on functional outcome in patients with anterior circulation ischaemic stroke having endovascular thrombectomy versus standard care: a meta-analysis of individual patient data. Lancet Neurol. 2018 Jan;17(1):47-53. doi: 10.1016/S1474-4422(17)30407-6. Epub 2017 Dec 16. PMID 29263006
- [Result] Bouslama M, Haussen DC, Aghaebrahim A, Grossberg JA, Walker G, Rangaraju S, Horev A, Frankel MR, Nogueira RG, Jovin TG, Jadhav AP. Predictors of Good Outcome After Endovascular Therapy for Vertebrobasilar Occlusion Stroke. Stroke. 2017 Dec;48(12):3252-3257. doi: 10.1161/STROKEAHA.117.018270. Epub 2017 Oct 31. PMID 29089457
- [Result] Terceno M, Silva Y, Bashir S, Vera-Monge VA, Cardona P, Molina C, Chamorro A, de la Ossa NP, Hernandez-Perez M, Werner M, Camps-Renom P, Rodriguez-Campello A, Canovas D, Purroy F, Serena J; Catalan Stroke Code and Reperfusion Consortium (Cat-SCR). Impact of general anesthesia on posterior circulation large vessel occlusions after endovascular thrombectomy. Int J Stroke. 2021 Oct;16(7):792-797. doi: 10.1177/1747493020976247. Epub 2020 Dec 1. PMID 33573525
- [Result] Gory B, Mazighi M, Labreuche J, Blanc R, Piotin M, Turjman F, Lapergue B; ETIS (Endovascular Treatment in Ischemic Stroke) Investigators. Predictors for Mortality after Mechanical Thrombectomy of Acute Basilar Artery Occlusion. Cerebrovasc Dis. 2018;45(1-2):61-67. doi: 10.1159/000486690. Epub 2018 Jan 30. PMID 29393092
- [Result] Schonenberger S, Henden PL, Simonsen CZ, Uhlmann L, Klose C, Pfaff JAR, Yoo AJ, Sorensen LH, Ringleb PA, Wick W, Kieser M, Mohlenbruch MA, Rasmussen M, Rentzos A, Bosel J. Association of General Anesthesia vs Procedural Sedation With Functional Outcome Among Patients With Acute Ischemic Stroke Undergoing Thrombectomy: A Systematic Review and Meta-analysis. JAMA. 2019 Oct 1;322(13):1283-1293. doi: 10.1001/jama.2019.11455. PMID 31573636
- [Result] Cappellari M, Pracucci G, Forlivesi S, Saia V, Nappini S, Nencini P, Inzitari D, Greco L, Sallustio F, Vallone S, Bigliardi G, Zini A, Pitrone A, Grillo F, Musolino R, Bracco S, Tinturini R, Tassi R, Bergui M, Cerrato P, Saletti A, De Vito A, Casetta I, Gasparotti R, Magoni M, Castellan L, Malfatto L, Menozzi R, Scoditti U, Causin F, Baracchini C, Puglielli E, Casalena A, Ruggiero M, Malatesta E, Comelli C, Chianale G, Lauretti DL, Mancuso M, Lafe E, Cavallini A, Cavasin N, Critelli A, Ciceri EFM, Bonetti B, Chiumarulo L, Petruzzelli M, Giorgianni A, Versino M, Ganimede MP, Tinelli A, Auteri W, Petrone A, Guidetti G, Nicolini E, Allegretti L, Tassinari T, Filauri P, Sacco S, Pavia M, Invernizzi P, Nuzzi NP, Carmela Spinelli M, Amista P, Russo M, Ferrandi D, Corraine S, Craparo G, Mannino M, Simonetti L, Toni D, Mangiafico S. General Anesthesia Versus Conscious Sedation and Local Anesthesia During Thrombectomy for Acute Ischemic Stroke. Stroke. 2020 Jul;51(7):2036-2044. doi: 10.1161/STROKEAHA.120.028963. Epub 2020 Jun 10. PMID 32517584
- [Result] Butt W, Dhillon PS, Podlasek A, Malik L, Nair S, Hewson D, England TJ, Lenthall R, McConachie N. Local anesthesia as a distinct comparator versus conscious sedation and general anesthesia in endovascular stroke treatment: a systematic review and meta-analysis. J Neurointerv Surg. 2022 Mar;14(3):221-226. doi: 10.1136/neurintsurg-2021-017360. Epub 2021 Mar 23. PMID 33758063
- [Result] Brinjikji W, Pasternak J, Murad MH, Cloft HJ, Welch TL, Kallmes DF, Rabinstein AA. Anesthesia-Related Outcomes for Endovascular Stroke Revascularization: A Systematic Review and Meta-Analysis. Stroke. 2017 Oct;48(10):2784-2791. doi: 10.1161/STROKEAHA.117.017786. Epub 2017 Sep 13. PMID 28904228